CLINICAL TRIAL: NCT05273762
Title: Treatment of Low-Risk Submassive Pulmonary Embolism With FlowTriever: Efficacy and Safety
Brief Title: Treatment of Low-Risk Submassive Pulmonary Embolism With FlowTriever
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-1117
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FlowTriever (Experimental)
  Interventions: Device: FlowTriever

INTERVENTIONS:
Device: FlowTriever — Mechanical thrombectomy for pulmonary embolism

SUMMARY:
This study is focused on investigating the efficacy and safety of the FlowTriever device to treat low-risk submassive pulmonary embolism.

DETAILED DESCRIPTION:
In this study, patients that present with low-risk submassive pulmonary embolism with hemodynamic stability and with either positivity of cardiac biomarkers, or radiographic or echocardiographic evidence of right ventricular strain will be assigned to be treated with mechanical thrombectomy, which includes conscious sedation, via FlowTriever.

ELIGIBILITY:
INCLUSION CRITERIA

I1. ≥ 18 years of age

I2. Clinical signs and symptoms of low-risk Intermediate pulmonary embolism defined per 2019 ESC Guidelines:

Only one of the following:

* Presence of either RV strain or RV dilation on CT scan or Echo TTE
* 4th generation Troponin T > 0.01 ng/mL or 5th generation Troponin T >14 ng/L

Troponin I > 51.4 ng/L (Northwell reference laboratory)

I3. sPESI score 0 or >1*

*Signs of RV dysfunction on Echo TTE or CTPA or elevated cardiac biomarker levels may be present, despite a calculation of sPESI 0.

I4. Echocardiogram, Computed Tomography Pulmonary Angiogram, or pulmonary angiographic evidence of proximal filing defect in at least one main, lobar, or segmental pulmonary artery with or without pulmonary infarction

I5. Hemodynamically stable

EXCLUSION CRITERIA

E1. Patients with active and severe COVID-19 infection (e.g. using ventilator, requiring hemodynamic support)

E2. Unable to anti-coagulate with heparin or alternative

E3. Known sensitivity to radiographic contrast agents that cannot be pre-treated

E4. Life expectancy < 6 months

E5. Current participation in another study that may interfere with the patient's participation in this study.

E6. Inability to consent

E7. Patient is pregnant or plans to become pregnant within the next 6 months and/or currently breastfeeding.

E8. Subsegmental pulmonary embolism only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in mMRC dyspnea score from | Baseline (state at time of admission to hospital) to 30-day follow-up.

SECONDARY OUTCOMES:
Change in Pulmonary Embolism Quality of Life Questionnaire (PEmbQOL) | Procedure to 30-day, 3-month, and 6-month follow up.
Change in Six Minute Walk Test (6MWT) (distance covered in meters over 6 minutes) | Pre-procedure to 30-day, 3-month, and 6-month follow up.
Echocardiogram Measurements: Change | Pre-procedure to 30-day and 6-month follow up
Echocardiogram Measurements: Change | From pre-procedure echocardiogram compared to 30-day and compared to 6-month follow up
ICU Length of Stay | Length of index hospitalization, length of hospitalization median of 9.1 days, length of ICU stay median 3.1 per JNS
  Time spent in the Intensive Care Unit (ICU) for the length of the hospital visit.
Hospital Duration | Length of index hospitalization, length median of 9.1 days per AHA journal
Device related death Device related bleeding Device related vascular injury Device related cardiac injury Clinical deterioration Rescue intervention | From end of index hospitalization to 30 days post-procedure, whichever comes first
Change in hemodynamic measurements | Before insertion of device during the procedure compared to 5 minutes after device is removed
Site Complications | Length of index hospitalization, length median of 9.1 days per AHA journal
Oxygen Requirement | Length of index hospitalization, length median of 9.1 days per AHA journal
All-cause Mortality | Length of index hospitalization, length median of 9.1 days per AHA journal
Bleeding Re-thrombosis Edema Pain | From end of index hospitalization to 30 days post-procedure, whichever comes first

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northern Westchester Hospital, Mount Kisco, New York
  - Lenox Hill Hospital, New York, New York